CLINICAL TRIAL: NCT07245160
Title: Feasibility Study of Addressing Anxiety in Children With ASD and Intellectual Disability Through the Facing Your Fears Program
Brief Title: A Cognitive Behavioral Therapy Approach to Addressing Anxiety in Children With ASD and Intellectual Disability
Acronym: FYF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Janys Lim, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSREB #124721
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder (ASD); Intellectual Disability
Keywords: autism spectrum disorder; ASD; anxiety; cognitive behavioral therapy; intellectual disability
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Intervention (Experimental): The experimental condition is a cognitive behavioral therapy intervention that is typically geared for children with ASD without intellectual disability. The established CBT, Facing Your Fears, supports participants in the following key areas: 1) building emotional regulation, 2) developing cognitive tools such as positive self-talk and affirmations, 3) enhancing coping strategies adapted to individual sensory and regulatory profiles, and 4) engaging in gradual exposure to situations or stimuli. The experimental condition will apply the Facing Your Fears model to children with ASD and intellectual disability.
  Interventions: Behavioral: Facing your Fears
- Wait-List Control (Other): A wait-list control design is employed to ethically evaluate the impact of a CBT intervention. Participants are initially screening using a comprehensive battery of standardized assessments to establish baseline functioning. The assessments include the SCARED/ MASC-2 to evaluate anxiety symptoms; CBCL to evaluate emotional behavioral problems; PedsQL to measure health-related quality of life; ADOS to support diagnostic clarity for autism spectrum characteristics; and the WASI to assess cognitive function and IQ. Following this pre-intervention phase, participants enter a wait-list control period where they do not receive the CBT intervention. The waiting period serves as the control condition, providing natural comparison for later outcomes. Once their cycle is assigned, the same participants transition into the experimental phase.
  Interventions: Behavioral: Baseline Treatment

INTERVENTIONS:
Behavioral: Facing your Fears — The Facing Your Fears intervention is a cognitive behavioral therapy program for children with ASD that is designed to establish somatic and emotional regulation strategies and enhance the use of personalized cognitive coping mantras through a gradual exposure to feared or anxiety provoking situations. The FYF program was developed for children with ASD, but prior research did not assess the feasibility of applying this intervention in children with ASD and intellectual disability. The intervention in the experimental condition will apply this core foundation of the FYF intervention to children with ASD and intellectual disability.
  Arms: Cognitive Behavioral Intervention
Behavioral: Baseline Treatment — The wait-list control condition is utilized as a baseline treatment phase where participants undergo a comprehensive battery of standardized assessments to establish baseline functioning. The SCARED/ MASC-2, CBCL and PedsQL is used to assess anxiety symptoms, identify co-occurring issues (e.g., aggression and attention problems) and overall well-being and functioning. Assessments such as the ADOS and WASI are semi-structured, direct observations, which confirm ASD diagnosis for study eligibility and estimates general cognitive ability and IQ. The results from these assessments will confirm eligibility for the study and provide baseline results for post-intervention analysis. The purpose of this pre-intervention phase is to establish a detailed baseline of each participant's functioning across key domains, provide diagnostic clarity and control for confounding variables (e.g., IQ), and enable analysis through pre and post comparison to assess the proposed intervention's effectiveness.
  Arms: Wait-List Control

SUMMARY:
Anxiety can be a debilitating and common concomitant diagnosis in autism spectrum disorders (ASD). Dependent on age and subtype of anxiety, the prevalence of anxiety in individuals with autism ranges between 1.7-84%. Meanwhile, the prevalence rate of intellectual disability (ID) in individuals with ASD ranges between 50-80% based on previous studies. There is an even greater risk of anxiety, ranging between 13.6- 43%, in individuals with ASD and ID. Despite the high prevalence of anxiety within this population, there are limited studies exploring assessments and treatments geared towards addressing anxiety in autism and intellectual disabilities. Previous studies have been limited to children who are identified as high functioning, or identified as low functioning without a concomitant diagnosis of ID. Given this, the present study focuses on the population of individuals with ASD and ID by exploring the feasibility of a CBT intervention designed for individuals with high-functioning autism

This pilot study aims at addressing and treating anxiety in children with ASD and intellectual disability through the Facing Your Fears (FYF) intervention. Facing Your Fears is a cognitive behavioral therapy (CBT) program specifically designed to address anxiety symptoms in children with autism. Research exploring the effectiveness of the FYF intervention within the population of individuals with ASD and ID is limited. This study aims at evaluating the feasibility of the Facing Your Fears program to address anxiety in children with ASD and ID, while evaluating the effectiveness of this intervention in larger group settings. The duration of the study will run over two 12-week cycles with study assessments conducted in-person, once a week. The study will involve 5-6 parent-child dyads to make up 10-12 participants per cycle. The child participants must be between the ages of 12-18 years old and have a confirmed diagnosis of ASD that meets DSM-V criteria. The study will commence with a month of recruitment, and a month allotted for collating data and assessments, before and after each 12-week intervention cycle. Evaluations will take place at screening, every study visit, and post intervention. Alongside the study evaluations, weekly sessions will involve didactic and practice sessions, with the last 30 minutes reserved for parent training. The sessions focus on the use and generalization of the taught strategies to address anxious symptoms, and exposure sessions outside of the weekly sessions. At the end of the 12-week cycle, the assessments related to the study outcomes will be administered again to allow investigators to compare and analyze pre- and post-intervention scores.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental condition that is characterized by social communication deficits and restricted and repetitive behaviours. Its prevalence is estimated at 1 in every 59 children or 1-2% of the population in Asia, Europe, and North America. There are about four males for every female who receives the diagnosis. While the exact cause is still unknown, it is postulated that it may be due to a combination of genetics, environmental, and epigenetic factors. There are a number of other disorders that are associated with autism spectrum disorder, such as intellectual disability, anxiety, Fragile X, and ADHD. Of these co-morbid conditions, anxiety is one of the most prevalent comorbid psychiatric problems in children with autism. Prevalence rates of anxiety in individuals with autism range between 1.7-84%, depending on age and subtype of anxiety. Meanwhile, prevalence range of intellectual disability in individuals with autism ranges between 50-80% based on previous studies. In individuals with autism and intellectual disability, there is an even greater risk of anxiety, ranging between 13.6-43%.

However, despite the high prevalence rate of anxiety within this population, there are not a lot of studies that have looked into assessments and treatment for individuals with autism and intellectual disabilities. Most studies on anxiety in autism have been in individuals without a concomitant diagnosis of intellectual disability. Only two reviews have previously evaluated therapy for anxiety in low-functioning individuals with autism, without "low-functioning" being equivalent to a diagnosis of intellectual disability. In fact, a lot of individuals with intellectual disabilities are usually found ineligible to be part of studies as a lot of assessments in these studies rely on self-reports of internal states. Limitations of cognition and communication skills may make reliability of responses to assessments challenging. Thus, while there are some interventions available to individuals with autism and intellectual disability to address their anxiety, to our knowledge, there are no studies that have looked into evaluating the effectiveness of these interventions in larger groups. There are also no studies that have looked into the feasibility of using existing interventions for addressing anxiety in autism, in children with autism and intellectual disability. Facing Your Fears program is a cognitive behavioural therapy (CBT) program specifically designed for children with autism who are experiencing anxiety. However, previous studies have been limited to children who are identified as high functioning autism. This will be a feasibility study on the use of the Facing Your Fears program in addressing anxiety in children with autism and intellectual disability.

Potential participants will be invited to join the study through assigned research staff who will introduce the study, the Facing Your Fears program, and assessed for eligibility. Once they are deemed eligible and express interest, they will be invited to come in for an appointment to discuss and sign consent and assent forms. Once the consent and assent forms are signed, the guardian will be interviewed by an assigned research staff following a screening interview. The screening and baseline phase will include a structured interview regarding the participant's medical history, and standardized questionnaires and assessments. These assessments will include:

1. SCARED/MASC-2 (parent and child report forms for anxiety symptoms)
2. CBCL (parent-reported scale used as a screening measure for internalizing and externalizing behaviours of a child (preschool and school-age), which includes measures of social deficits. CBCL subtests include anxious/depressed, withdrawn, social problems, thought problems, attention problems, somatic complaints, and aggressive and/or delinquent behaviours)
3. ADOS (standardized play assessment for autism diagnosis)
4. WASI (Weschler Abbreviated Scale for Intelligence)
5. PedsQL (brief measure of health-related quality of life in children and young people composed of generic core scales: physical functioning, emotional functioning, social functioning, and school functioning)
6. Satisfaction Questionnaire (only administered post the 12 week period) Participants who meet eligibility criteria based on inclusion/exclusion criteria will be enrolled in the study. Those who do not meet criteria will be considered a screen fail.

Following the screening/baseline period, eligible participants will be assigned to treatment groups of 5-6 child-parent dyads who will meet once a week for 1.5 hours, over a 12-week period (N=24; 12 participants per cycle). Participants will be assigned to the cycles based on the order in which they are screened and enrolled. The first 6 parent-child dyads deemed eligible will begin treatment in cycle 1. The remaining 6 parent-child dyads deemed eligible will begin treatment in cycle 2. These weekly sessions will be a combination of didactic and practice sessions, with the last 30 minutes reserved for parent training. Participants will be provided a schedule of sessions to attend. Facing Your Fears workbooks for both parent and child will be provided for use during the sessions. Assessment forms and questionnaires will also be provided for the parent to answer during this visit.

1. SCARED/MASC-2
2. CBCL
3. PedsQL

The initial session includes the introduction to anxiety, signs and symptoms, situations that can cause anxiety, and an introduction to some strategies to address anxiety. The program focuses on the use and generalization of the strategies in the sessions to address anxious symptoms, and exposure sessions outside of the sessions.

The same guardian will accompany the participant to every session to learn about anxiety disorders and the basic principles of CBT. The guardian helps identify the specific anxiety symptom of the participant to target during the study, discussion of guardian's own concerns, and the challenges in managing anxiety in the context of ASD and intellectual disability. The sessions will follow the flow set out in the Facing Your Fears workbooks as this program was specifically designed for children with autism.

At the end of the 12-week period, the MASC-2/SCARED, PedsQL, CBCL, and Satisfaction Questionnaire will be administered again. Pre- and post-intervention scores will be collected and analyzed. Outcomes of the post-intervention assessments will undergo t-test analysis comparing pre and post test results of study measures to determine statistically significant change after exposure to the intervention. The change in proportion of the participants whose scores met clinical cut-off T-scores will also be determined, by comparing pre and post intervention scores on study measures. Surveys will be completed by participant dyads to assess for the feasibility of the intervention's recruitment, intensity, frequency, and duration of the modified intervention for this new target population. The preliminary responses of the participants to the intervention will also be assessed. The study team will be analyzing if the data collection procedures and outcome measures are feasible and appropriate. A survey will also be completed by facilitators in order to determine whether the intervention and study procedures are acceptable, as well as determine potential areas of concern during implementation. Cost analyses of the study will also be completed during and at the end of the study.

This study will be asking participants and their parents to talk about their worries and fears. Talking about these topics and the gradual exposure to challenge their fears may cause distress and discomfort. To mitigate distress experienced, should the participants feel that the rate of exposure is causing too much distress, the rate of exposure may be individualized for the participants. Participants will be monitored throughout the study by the facilitators to determine possible adverse events' onset, relation to study intervention, and outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 12-18 years
2. Confirmed diagnosis of ASD that meets DSM-V criteria
3. ADOS scores consistent with an ASD diagnosis
4. WASI scores equivalent to 50-70
5. CBCL with T score >/= 70 for the anxiety subscale
6. MASC-2/SCARED score with T-scores reflecting clinically significant anxiety
7. Not part of another interventional study or clinical trial
8. Stable non-pharmacological therapies for at least 12 weeks
9. Stable pharmacological therapies for at least 8 weeks
10. Will not start new treatment for anxiety, medication or intervention, within the study 12 week study period
11. Consistent parent partner per child throughout the duration of the study

Exclusion Criteria:

1. Individuals with history of significant suicidal ideations or attempts
2. Individuals involved in a concurrent interventional study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in score on the Screen for Child Anxiety Related Disorders (SCARED) | SCARED will be administered at screening, at Week 6, and then at Week 12.
  The SCARED is a 41-item child and parent reported questionnaire that assesses anxiety disorders in childhood and adolescence. A total score on each scale of 25 or higher may indicate the presence of an anxiety disorder. The items reflect domains of anxiety such as panic disorder, generalized anxiety disorder, separation anxiety disorder, social anxiety disorder and school avoidance. For example, a score of 3 for items 11, 17, 36 may indicate significant school avoidance. Pre and post intervention scores (i.e., total and domain specific) will be compared for clinical significance. A lower total score post-intervention may indicate improvement or reduction in anxiety symptoms. A drop of 5-10 points or more in total score may be clinically meaningful, depending on baseline severity. Changes in scores within the domains reflect how specific anxiety symptoms have responded to intervention. Lower domain scores post-intervention would suggest a positive change within that domain.
Changes in Multidimensional Anxiety Scale for Children | Second Edition (MASC-2) score | MASC-2 test retest intervals are 3 weeks- 3 months. The assessment will be administered at screening and at the end of the study (Week 12).
  The MASC-2 is a 50-item child and parent reported questionnaire that assesses the presence of symptoms related to anxiety disorders in domains such as separation and social anxiety, general anxiety disorder, harm avoidance, obsessions and compulsions and physical symptoms. Raw scores for each item are converted to T-scores, percentiles and confidence intervals. Elevated T-scores in one or more domains suggest which type of anxiety is likely prominent. The scale will be administered pre-intervention, during intervention and post-intervention. A lower score post-intervention may indicate an improvement or reduction in anxiety symptoms. Lower total T-scores suggest a general decrease in overall anxiety symptoms compared to baseline. Lower subscale scores (e.g., Social Anxiety, Separation Anxiety, etc.) suggest a symptom reduction in the specific domains. A lower score may not mean full remission, but significant symptom relief (e.g., improved functionality and emotional regulation).

SECONDARY OUTCOMES:
Changes in the Child Behavior Checklist (CBCL) scores. | CBCL has a test-retest interval of 6 months. The measure will be done at screening, EOS (week 12) and post-intervention (Week 24).
  The Child Behavior Checklist (CBCL) school-aged version (6-18 years old) is a parent-reported scale assessing a wide range of emotional and behavioral problems in children and adolescents. CBCL subtests include anxious/depressed, withdrawn, social problems, thought problems, attention problems, somatic complaints, and aggressive and/or delinquent behaviors. The response scale includes 3 items, 0= not true, 1=somewhat or sometimes true, 2= very or often true, making up the raw score. The raw score is converted to standardized T-scores using age- and gender-specific norms. Normal range correlates to a T-Score of <65, borderline clinical correlates to a T-Score of 65-69, and a clinical range correlates to a T-Score of 70 or higher. A decrease in T-Score in post-intervention compared to pre-intervention would suggest a likely clinical improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital- LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The results will be published collectively, and we will not be sharing individual participant data.

REFERENCES:
- [Background] Reaven J, Blakeley-Smith A, Leuthe E, Moody E, Hepburn S. Facing your fears in adolescence: cognitive-behavioral therapy for high-functioning autism spectrum disorders and anxiety. Autism Res Treat. 2012;2012:423905. doi: 10.1155/2012/423905. Epub 2012 Oct 3. PMID 23091719